CLINICAL TRIAL: NCT06504745
Title: The Effect of Peer Education on the Knowledge and Skill Levels of Nursing Students in Physical Evaluation of the Newborn: A Pre/Post-test Comparative Study
Brief Title: The Effect of Peer Education on the Knowledge and Skill Levels of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Signem ANOL KILIÇ, research assistant, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 255515
Record Dates: First submitted 2024-06-25; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Students; Nursing
Keywords: peer education; nursing education; newborn physical examination; nursing practice
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Intervention group: peer education Control group: instruction education
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Peer educator students group (a group of six senior nursing students), provided Newborn Physical Assessment training to 4th-year students in the nursing laboratory every week. Each training was conducted with a group of 5 students. This each training consisted of 30 minutes of theoretical presentation using a PowerPoint presentation material and 20 minutes of skills application on a newborn model, totaling 50 minutes. Before the training, the NPA-KT was administered, and the students' skills were evaluated using the NPA-SCL. At the end of the training, the NPA-KT and the Peer Support Scale were administered to the students. Three weeks after the training, the students' knowledge levels were re-evaluated using the NPA-KT.
  Interventions: Other: Peer education
- Control Group (Active Comparator): The researchers provided Newborn Physical Assessment training to 4th-year students in the nursing laboratory every week. Each training was conducted with a group of 5 students. This training consisted of 30 minutes of theoretical presentation using a PowerPoint presentation material and 20 minutes of skills application on a newborn model, totaling 50 minutes. Before the training, the NPA-KT was administered, and the students' skills were evaluated using the NPA-SCL. At the end of the training, the NPA-KT and the Peer Support Scale were administered to the students. Three weeks after the training, the students' knowledge levels were re-evaluated using the NPA-KT.
  Interventions: Other: control group

INTERVENTIONS:
Other: Peer education — experimental group
  Arms: Intervention Group
Other: control group — instruction training
  Other Names: instruction training
  Arms: Control Group

SUMMARY:
This study was planned to determine the impact of peer education and instruction received from the instructor on the knowledge and skill levels of students in the physical assessment of the newborn.

DETAILED DESCRIPTION:
Nursing education is a process that involves the transfer of theoretical knowledge, skills, and attitudes based on cognitive, affective, and psychomotor domains into clinical practice.The aim is to train nurses who are capable of evidence-based intervention in line with holistic care principles in clinical settings. However, the process of transferring theoretical knowledge and skills acquired by students into clinical practices takes place in complex social environments in clinics, unlike traditional classroom settings.

Among student-centered teaching methods, 'peer education' has gained considerable attention in recent years. If peer-to-peer education can attain similar learning outcomes as standard teaching methods, it is believed that it can be applied to learning objectives encompassing many professional knowledge and skill techniques.

Physical examination of the newborn requires considerable knowledge, skill and experience.

This situation is known to impose limitations on nursing students in applying and learning newborn care based on atraumatic care principles in clinical settings. Additionally, the fear of causing harm to the newborn or inflicting pain experienced by nursing students creates emotional and mental stress situations, making it difficult for the instructor to teach and reinforce care practices in newborn nursing.

Therefore, this study was planned to compare the difference between peer educators and instructors in the physical examination of newborns in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Volunteer to participate in the study
* 4th-year nursing students

Exclusion Criteria:

* Non-volunteering

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
The Newborn Physical Assessment Skills Control List (NPA-SCL) | In this study, the skill level of the students was measured at the time of application in the laboratory after the training after the training in 1 hour.
  NPA-SCL includes the measurement and evaluation of a newborn's height, weight, head circumference, chest circumference, and abdominal circumference. objectively evaluate the student during the laboratory practice conducted in the study, the NPA-SCL was prepared by the responsible researchers based on the literature. In the evaluation of the Control List, the student is expected to evaluate each item as 'Not Applied=0 points', 'Partially Applied=1 point', and 'Applied=2 points' according to their performance. The minimum score a student can receive from the Control List is 0 points and the maximum is 46 points. After the form was prepared by the researchers, it was presented to 6 experts. Based on expert opinions, the form was finalized.
The Newborn Physical Assessment Knowledge Test (NPA-KT) | In the study, knowledge level of the students was measured with pre-test (before the training), post-test 1 (after the training in one hour), and post-test 2 (3 weeks later)
  This form, prepared by researchers based on the literature, consists of 20 questions. Each question is worth 5 points. Participants are expected to answer each item on the knowledge test as 'Correct', 'Incorrect', or 'Don't know'. Scores on the knowledge test range from a minimum of '0 points' to a maximum of '100 points'. After the form was prepared by the researchers, it was presented to 3 faculty members from the Department of Fundamentals of Nursing and 3 faculty members from the Department of Child Health and Diseases Nursing for their opinions. Based on their expert opinion, the form was finalized

SECONDARY OUTCOMES:
Peer Support Scale (PSS) | Within one hour after the training was completed, only the peer support level of the intervention group was measured.
  The Peer Support Scale was developed by Kuo et al. in 2007 to measure nursing students' collaboration with each other. The scale consists of a total of 17 items, comprising three subscales: physical support, academic support, and emotional support. The overall score of the scale provides the score for nursing students' collaborative behaviors with each other. All items on the scale are positively phrased and rated on a 4-point Likert scale: Disagree (1), Partially Disagree (2), Agree (3), Completely Agree (4). In the study

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I want to share my research protocol after one year.

REFERENCES:
- [Background] Fard ZR, Azadi A, Khorshidi A, Mozafari M, O'Connor T, Budri AMV, Moore Z, Patton D. A comparison of faculty led, mentorship program and peer mentoring on nursing students wound dressing clinical skills. Nurse Educ Today. 2020 Jun;89:104378. doi: 10.1016/j.nedt.2020.104378. Epub 2020 Feb 19. PMID 32209490
- [Result] Kuo CL, Turton MA, Lee-Hsieh J, Tseng HF, Hsu CL. Measuring peer caring behaviors of nursing students: scale development. Int J Nurs Stud. 2007 Jan;44(1):105-14. doi: 10.1016/j.ijnurstu.2006.07.025. Epub 2006 Oct 6. PMID 17027986
- [Result] Joung J, Kang KI, Yoon H, Lee J, Lim H, Cho D, Cha M, Choi B. Peer mentoring experiences of nursing students based on the caring perspective: A qualitative study. Nurse Educ Today. 2020 Nov;94:104586. doi: 10.1016/j.nedt.2020.104586. Epub 2020 Aug 29. PMID 32932060